CLINICAL TRIAL: NCT07254845
Title: A PROSPECTIVE, SINGLE-CENTERED, ASSESSOR-BLINDED STUDY TO EVALUATE THE CLINICAL EFFICACY OF THE PROPOSED CELL/TISSUE HISTOPATHOLOGY PROCESSOR CCELL (CONFOCAL FLUORESCENCE ENDOMICROSCOPY) FOR INTRAOPERATIVE DIAGNOSIS IN BRAIN TUMORS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VPIX Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: cCeLL_II_2025_Cedars
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Frozen Sections; Indocyanine Green (ICG); Brain Tumor
Keywords: diagnostic imaging; intraoperative; confocal laser endomicroscopy
MeSH Terms: conditions — Brain Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This prospective, multicenter, evaluator-blinded clinical trial evaluates the cCeLL - In vivo confocal laser fluorescence microscope for brain tumor diagnosis during surgery.
  Intervention Summary Study Type: Interventional (Diagnostic) Design: Single-group assignment, evaluator-blinded
  Intervention:
  1. ICG injection during surgery
  2. Fluorescence imaging of the tumor margin using cCeLL - In vivo
  3. Comparison with standard frozen and permanent section analyses
  4. Blinded evaluation by pathologists This study aims to enhance tumor margin assessment and improve diagnostic accuracy during brain tumor surgery.
Masking Description: Pathologists will perform diagnoses without access to patient medical records and will not see prior diagnostic results. They will assess tissue samples using only de-identified information, ensuring that fluorescence imaging results do not influence their evaluation. This approach eliminates bias and maintains the integrity of the study's diagnostic comparison.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cCeLL - In vivo Imaging (Experimental): Participants diagnosed with brain tumors will receive an intravenous injection of Indocyanine Green (ICG) during surgery. The cCeLL - In vivo confocal laser fluorescence microscope will be used to capture real-time images of the tumor margins before tissue collection. Standard frozen section and permanent section analyses will then be performed for diagnostic comparison.
  Interventions: Device: cCeLL In vivo; Drug: Indocyanine Green

INTERVENTIONS:
Device: cCeLL In vivo — Dosage Form: Intravenous injection Dosage: 0.1 - 0.5 mg/kg of Indocyanine Green (ICG) Frequency: Single administration during surgery Duration: Real-time imaging performed immediately after ICG injection and used intraoperatively for tumor margin assessment
Drug: Indocyanine Green — fluorescence dye for staining tissue

SUMMARY:
The primary objective of this single-center study is to demonstrate the performance of cCeLL, used in real time, compared to frozen section analysis. The investigational device is intended for use with indocyanine green (ICG) for fluorescence imaging as an aid in the visualization of vessels (micro- and macro-vasculature) blood flow in the cerebrovascular before, during or after cranial diagnostic and therapeutic procedures, such as tumor biopsy and resection, and the images will be immediately transmitted to a single pathologist for real-time evaluation, without influencing the surgical decision-making process. The comparison will be made between the device and the conventional intraoperative histological frozen section analysis of identical brain tissue samples in the same patient. Both methods will be compared in terms of their accuracy using the standard of practice, the final pathological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older as of the screening date
2. Patients suspected of having a brain tumor who are scheduled for neurosurgery and are considered candidates for tumor resection
3. Patients who understand and have signed the informed consent form

Exclusion Criteria:

1. Specimens obtained from patients who have agreed to participate in this clinical trial and who meet the inclusion criteria
2. Normal tissue specimens obtained unavoidably during tumor resection surgery in tumor patients
3. Tissue samples must be adequate for both FS and PS analysis
4. Minimum lesion size of 1 cm for reliable cCeLL imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of cCeLL imaging, compared with frozen section (FS), using the permanent section (PS) as the reference standard. | Visit 1 (Surgery Day / Intervention Day) as D-Day
  cCeLL and FS diagnostic accuracy will be compared to PS, reporting sensitivity, specificity, PPV, NPV, and overall accuracy with 95% CIs. Analyses are descriptive, summarized by dataset, tumor type, and sampling site.

SECONDARY OUTCOMES:
Diagnostic Performance of cCeLL vs FS Across Tumor Types and Sampling Sites | Visit 1 (Surgery Day / Intervention Day) as D-Day
  Diagnostic indices (sensitivity, specificity, accuracy) will be calculated for each tumor type and sampling site using PS as the reference.
  cCeLL and FS performance will be compared side by side within subgroups descriptively, without statistical testing due to small sample sizes.
Rate of Non-diagnostic Images with cCeLL | Visit 1 (Surgery Day / Intervention Day) as D-Day
  The number of non-diagnostic cCeLL images will be reported, with N_ND representing non-diagnostic images and N_Total the total images acquired.
Diagnostic Time Comparison (cCeLL vs FS) | Visit 1 (Surgery Day / Intervention Day) as D-Day
  Acquisition and interpretation times for cCeLL and FS will be summarized, with differences described; a positive value indicates time saved using cCeLL.
Time Required for cCeLL Imaging/Interpretation | Visit 1 (Surgery Day / Intervention Day) as D-Day
  The average and range of regions imaged per case, along with cCeLL acquisition and interpretation times, will be summarized to assess operational feasibility and real-time workflow integration during neurosurgery.
Detection of Positive Surgical Margins with cCeLL | Visit 1 (Surgery Day / Intervention Day) as D-Day
  For post-resection scans, biopsies will be performed only if cCeLL is positive, and the Positive Margin Detection Rate will be used to assess cCeLL's ability to identify residual tumor at surgical margins

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) may not be shared due to patient privacy concerns, confidentiality agreements, regulatory restrictions, ethical considerations, and institutional policies. Additionally, data protection laws (e.g., GDPR, HIPAA) and proprietary research interests may limit data availability to ensure compliance and safeguard participant information.